CLINICAL TRIAL: NCT01270581
Title: High Flow Nasal Cannula vs Bubble Nasal CPAP for the Treatment of Transient Tachypnea of the Newborn in Infants ≥ 35 Weeks Gestation
Brief Title: High Flow Nasal Cannula Versus Bubble Nasal CPAP for the Treatment of Transient Tachypnea of the Newborn in Infants ≥ 35 Weeks Gestation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of sufficient enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0603
Record Dates: First submitted 2010-12-21; First posted 2011-01-05 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: transient tachypnea of the newborn; high flow nasal cannula; bubble nasal; continuous positive airway pressure
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Flow Nasal Cannula (Experimental): Unlike the nasal prongs for NCPAP (which fit tightly in the nares), the nasal cannula for HFNC have smaller, loose-fitting prong. With HFNC, positive airway pressure is achieved by high gas flow through the cannula into the external nares which provide resistance to expiration and facilitate inspiration. The distending pressure is determined by the size and structure of the nasal cannula, gas flow rate, and the neonate's airway anatomy 4,5,7. Newborns randomized to HFNC will be started on a flow rate of 4L/min and supplemental oxygen will be provided to maintain oxygen saturations between 88-93% (experimental group). Once initiated, the gas flow rate will be titrated as needed by the attending neonatologist to ameliorate signs of respiratory distress to a maximum flow rate of 6L/min. The nasal cannula size (0.2 cm or 0.3 mm outer diameter) will determined by the caliber of the subject's nares).
  Interventions: Other: High Flow Nasal Cannula
- Control Group- Bubble Nasal CPAP (Active Comparator): NCPAP provides continuous distending airway pressure during inspiration and expiration via nasal prongs; this has been shown to increase lung volume by increasing alveolar size, recruiting collapsed alveoli, and preventing atelectasis. Improved lung volumes decrease V/Q mismatch and improve the clinical course of neonates with RDS, and as such, early NCPAP use often avoids the need for intubation and mechanical ventilation. Newborns receiving bubble NCPAP will be placed on a PEEP 5cm H2O, and supplemental oxygen will be provided to maintain oxygen saturation between 88-93% (standard of care group) as is standard practice. The size of the nasal prongs used will be based on the subject's weight as per the manufacturer instructions.
  Interventions: Other: Bubble Nasal CPAP

INTERVENTIONS:
Other: High Flow Nasal Cannula — Humidified high flow nasal cannula (HFNC) has emerged as an alternative respiratory modality for late preterm newborns with respiratory distress. Like NCPAP, oxygen is delivered to the infant via nasal prongs and provides a continuous distending pressure. Unlike the nasal prongs for NCPAP (which fit tightly in the nares), the nasal cannula for HFNC have smaller, loose-fitting prong. With HFNC, positive airway pressure is achieved by high gas flow through the cannula into the external nares which provide resistance to expiration and facilitate inspiration. The distending pressure is determined by the size and structure of the nasal cannula, gas flow rate, and the neonate's airway anatomy 4,5,7.
  Arms: High Flow Nasal Cannula
Other: Bubble Nasal CPAP — NCPAP provides continuous distending airway pressure during inspiration and expiration via nasal prongs; this has been shown to increase lung volume by increasing alveolar size, recruiting collapsed alveoli, and preventing atelectasis. Improved lung volumes decrease V/Q mismatch and improve the clinical course of neonates with RDS, and as such, early NCPAP use often avoids the need for intubation and mechanical ventilation. Newborns receiving bubble NCPAP will be placed on a PEEP 5cm H2O, and supplemental oxygen will be provided to maintain oxygen saturation between 88-93% (standard of care group) as is standard practice. The size of the nasal prongs used will be based on the subject's weight as per the manufacturer instructions.
  Arms: Control Group- Bubble Nasal CPAP

SUMMARY:
The primary objective is to determine whether High Flow Nasal Cannula (HFNC) is a superior respiratory modality for neonates ≥36 weeks with transient tachypnea of the newborn (TTN) when compared to the standard of care modality (NCPAP).

DETAILED DESCRIPTION:
Transient Tachypnea of the Newborn, fetal lung fluid retention causing poor lung compliance and atelectasis, is a common entity in neonates ≥ 36 weeks in our unit. Currently our standard of care includes using the respiratory modality of bubble nasal continuous positive airway pressure (BNCPAP) to support these neonates during this illness. BNCPAP provides positive distending pressure to recruit alveoli and prevent atelectasis, however, it is associated with air leak (pneumothorax, pneumomediastinum), nasal irritation and necrosis, and intolerance. HFNC is another respiratory modality that uses high flow gas that also provides positive distending pressure and thus prevents atelectasis. This modality does not cause nasal irritation or necrosis and has a minimal risk of air leak. We postulate that HFNC is a superior modality to BNCPAP in treating neonates ≥ 36 weeks with TTN. This will be determined by comparing the duration of respiratory support (in hours) for newborns ≥ 36 weeks gestation with a diagnosis to TTN randomized to receive either NCPAP or HFNC for respiratory care.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 35 weeks
* diagnosis of TTN, defined as respiratory rate >60, presence of subcostal and /or intercostal retractions, nasal flaring, grunting, oxygen saturations 70-93% on room air, and radiological evidence of perihilar streaking and patchy infiltrates
* admission to the NICU at Mount Sinai hospital within first 24 hours of life

Exclusion Criteria:

* gestational age < 35 weeks
* history of thick meconium stained fluid and/or diagnosis of meconium aspiration syndrome
* diagnosis of major congenital pulmonary or cardiac anomalies
* initial CXR demonstrating air leak
* respiratory distress first occurring after 24 hours of life
* presumptive diagnosis of RDS as indicated by the need for FiO2 > 40%, severe retractions and grunting with poor air entry, and diffuse alveolar consolidation on chest radiograph

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Weintraub, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Dani C, Pratesi S, Migliori C, Bertini G. High flow nasal cannula therapy as respiratory support in the preterm infant. Pediatr Pulmonol. 2009 Jul;44(7):629-34. doi: 10.1002/ppul.21051. PMID 19499590
- [Background] Jasin LR, Kern S, Thompson S, Walter C, Rone JM, Yohannan MD. Subcutaneous scalp emphysema, pneumo-orbitis and pneumocephalus in a neonate on high humidity high flow nasal cannula. J Perinatol. 2008 Nov;28(11):779-81. doi: 10.1038/jp.2008.99. PMID 18974751
- [Background] Lampland AL, Plumm B, Meyers PA, Worwa CT, Mammel MC. Observational study of humidified high-flow nasal cannula compared with nasal continuous positive airway pressure. J Pediatr. 2009 Feb;154(2):177-82. doi: 10.1016/j.jpeds.2008.07.021. Epub 2008 Aug 30. PMID 18760803
- [Background] Locke RG, Wolfson MR, Shaffer TH, Rubenstein SD, Greenspan JS. Inadvertent administration of positive end-distending pressure during nasal cannula flow. Pediatrics. 1993 Jan;91(1):135-8. PMID 8416477
- [Background] Shoemaker MT, Pierce MR, Yoder BA, DiGeronimo RJ. High flow nasal cannula versus nasal CPAP for neonatal respiratory disease: a retrospective study. J Perinatol. 2007 Feb;27(2):85-91. doi: 10.1038/sj.jp.7211647. PMID 17262040
- [Background] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The NICU fellow on service, or on call, will identify all NICU admission that are potentially eligible for participation. Parents of potentially eligible subjects will be approached by a member of the NICU team to discuss study participation within 4 hours of admission to the NICU.
Period: Overall Study
Arm/Group | High Flow Nasal Cannula | Control Group- Bubble Nasal CPAP
Started | 4 | 3
Completed | 3 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Nasal Cannula | Control Group- Bubble Nasal CPAP | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Respiratory Support
Description: Data not collected due to insufficient enrollment for any data analysis.
Time Frame: average of 7 days
Arm/Group | High Flow Nasal Cannula | Control Group- Bubble Nasal CPAP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse event information not collected
Arm/Group | High Flow Nasal Cannula | Control Group- Bubble Nasal CPAP
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
low enrollment, data not analyzed - too small for any meaningful interpretation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes